CLINICAL TRIAL: NCT07134504
Title: Primary Diffuse Large B Cell Lymphoma (DLBCL) of the Prostate a Case Report
Brief Title: Primary Prostatic Lymphoma on a 66 Year-old Male in Mexico.
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, PHD, Instituto Mexicano del Seguro Social
Other Study IDs: 98207213
Record Dates: First submitted 2025-08-13; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: lymphoma; diffuse large B cell; urinary tract symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A 66-year-old male known case of diabetes and hypertension presented to the urology clinic with a 2-month history of lower urinary tract symptoms (LUTS), particularly poor flow, sense of incomplete bladder emptying, dysuria and hesitancy. Family history was negative for prostate or breast cancer.

On examination, there were signs of anaemia or lymphadenopathy. His abdominal examination was unremarkable with no hepatosplenomegaly, and his digital rectal examination (DRE) revealed an irregular, moderately enlarged nodular prostate.

DETAILED DESCRIPTION:
The patient underwent the following investigations in chronological order:

Laboratory investigations Haemoglobin: 134 g/L. Total leucocyte count: 8.6×109/L without any atypical cells. Platelets: 286×109/L. Prothrombin time/ International normalized ratio (PT/INR): 13/1.1. Creatinine: 1.1 mg/dL. Electrolytes: normal. Urine detailed report: normal. Urine culture and sensitivity: no bacterial growth. Prostate-specific antigen (PSA): 1.54 ng/mL. Radiological imaging Ultrasound of the kidney, ureter and bladder: normal non-hydronephrotic kidneys with 38 g prostate, with post void residual urine volume of 76 mL.

Based on suspicion of prostatic malignancy, he underwent MRI of the pelvis and lumbosacral (L/S) spine, whole body bone scan, and transrectal ultrasound (TRUS) guided 12-core needle biopsy of the prostate.

Bone scan: negative. MRI of the pelvis: 4.8×4.1×3.2 cm prostate with abnormal signal intensity area in the central zone appearing hypointense on T2-weighted image. The prostatic capsule and neurovascular bundles were intact.

Gross examination: TRUS biopsy showed 12 linear core tissues from both the right and left lobes of the prostate, with the largest measuring 1.1 cm.

Microscopic examination: sections from 4 cores out of 12 (2 each from the apical prostatic tissues of the right and left lobes) revealed prostate parenchyma infiltrated by atypical medium-sized to large-sized lymphoid cells arranged in diffuse sheets. These lymphoid cells exhibited scant to moderate amount of eosinophilic cytoplasm and nuclei with irregular contours, dispersed chromatin and occasional prominent nucleoli. The rest of the eight prostate tissue cores revealed benign prostate parenchyma showing glands lined by double-layered epithelium.

Immunohistochemical studies: tumour cells were strongly positive for leucocyte common antigen, CD20 (Pan-B marker), BCL-2 and CD10.The patient received alpha-adrenergic blocker tamsulosin with finasteride for LUTS with good response. For his radicular pain, he received diclofenac sodium and pregabalin. Following discussion in a multidisciplinary tumour board meeting, he received six cycles of R-CHOP (Rrituximab, Cyclophosphamide, Doxorubicin hydrochloride, Vincristine sulfate, and Prednisone) regimen at an outside cancer treatment facility.

ELIGIBILITY:
Inclusion Criteria:

- Patient with primary diffuse large B cell lymphoma

Exclusion Criteria:

* Patient with without primary diffuse large B cell lymphoma

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 66 Year old male.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
cancer specific survival | through the end of 6 cycles of R-CHOP an average of 6 months
  cancer specific survival with R-CHOP

CONTACTS AND LOCATIONS:
Locations (1):
- IMSS, Colonia del Valle, D.F, Mexico

IPD SHARING:
Plan to Share IPD: Yes
anyone who ask via e-mail
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: e-mail

REFERENCES:
- [Background] Bal S, Odujoko O, Fiedler J, Sieber SC, Beck E, Gupta G. Primary follicular lymphoma of the prostate co-existing with grade group 5 prostatic adenocarcinoma and presenting as a PI-RADS lesion 4 on mpMRI. Urol Case Rep. 2024 Mar 12;54:102708. doi: 10.1016/j.eucr.2024.102708. eCollection 2024 May. PMID 38550656